CLINICAL TRIAL: NCT02147990
Title: TIGER-2: A Phase 2, Open-label, Multicenter, Safety and Efficacy Study of Oral CO-1686 as 2nd Line EGFR-directed TKI in Patients With Mutant EGFR Non-small Cell Lung Cancer (NSCLC)
Brief Title: Multicenter Study of Rociletinib Administered to Patients With Previously Treated Mutant EGFR Non-small Cell Lung Cancer
Acronym: NSCLC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor discontinued development of CO-1686 for NSCLC.
Sponsor: Clovis Oncology, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO-1686-019 (TIGER-2)
Record Dates: First submitted 2014-05-13; First posted 2014-05-28 (Estimated); Results first posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-07

CONDITIONS: Non-small Cell Lung Cancer
Keywords: cancer; metastatic; locally advanced; lung; non-small cell lung cancer; NSCLC; epidermal growth factor receptor; EGFR; T790M; CO-1686; unresectable; recurrent; EGFR-directed therapy; irreversible EGFR inhibitor; TIGER; Rociletinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms; Neoplasm Metastasis; Recurrence | interventions — rociletinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rociletinib Mono-Therapy, T790M +ve (625mg BID) (Experimental): Starting dose of 625mg rociletinib, taken orally twice daily, with 8 oz (240 mL) of water and with a meal or within 30 minutes after a meal. Tablets should be swallowed whole. Treatment with rociletinib is continuous and each cycle will comprise of 28 days.
  Interventions: Drug: Rociletinib
- Rociletinib Mono-Therapy, T790M +ve (500mg BID) (Experimental): Starting dose of 500mg rociletinib, taken orally twice daily, with 8 oz (240 mL) of water and with a meal or within 30 minutes after a meal. Tablets should be swallowed whole. Treatment with rociletinib is continuous and each cycle will comprise of 28 days.
  Interventions: Drug: Rociletinib
- Rociletinib Mono-Therapy, T790M -ve (500mg BID) (Experimental): Starting dose of 500mg rociletinib, taken twice daily, with 8 oz (240 mL) of water and with a meal or within 30 minutes after a meal. Tablets should be swallowed whole. Treatment with rociletinib is continuous and each cycle will comprise of 28 days.
  Interventions: Drug: Rociletinib

INTERVENTIONS:
Drug: Rociletinib — Rociletinib will be administered to patients orally
  Other Names: CO-1686

SUMMARY:
The purpose of this study is to evaluate the safety and anti-tumor effect of rociletinib. The trial is open-ended, which means patients will continue to take rociletinib until the study doctor determines it is no longer beneficial for them.

DETAILED DESCRIPTION:
This is a Phase 2, single arm, open-label, dual cohort, multicenter study evaluating the safety and efficacy of rociletinib administered orally to patients with previously treated mutant EGFR NSCLC.

Patients will be enrolled into 2 cohorts. Cohort A will enroll approximately 125 eligible patients who are centrally confirmed T790M-positive. Cohort B will be a continuation of the study and will enroll up to approximately 100 eligible patients who will be either centrally confirmed T790M-positive or T790M-negative.

All patients (for Cohort A and B) should have experienced disease progression while on treatment with the first single-agent EGFR-directed TKI (EGFR-TKI) for advanced/metastatic NSCLC. One line of chemotherapy prior to the EGFR-TKI treatment is permissible.

The study (Cohorts A and B) will consist of a screening phase to establish study eligibility and document baseline measurements, an open-label treatment phase, in which the patient will receive rociletinib to ascertain safety and efficacy until disease progression as defined by RECIST Version 1.1, clinical tumor progression, or unacceptable toxicity as assessed by the investigator. For patients with clinical progression, radiographic assessment should be performed to document evidence of radiographic progression.

ELIGIBILITY:
Inclusion Criteria

* Histologically or cytologically confirmed metastatic or unresectable locally advanced NSCLC
* Documented evidence of a tumor with 1 or more EGFR mutations excluding exon 20 insertion
* Disease progression confirmed by radiologic assessment while receiving treatment with the first single agent EGFR-TKI
* EGFR TKI treatment discontinued less than or equal to 30 days prior to planned initiation of rociletinib
* The washout period for an EGFR inhibitor is a minimum of 3 days
* No intervening treatment between cessation of single agent EGFR TKI and planned initiation of rociletinib
* Previous treatment with less than or equal to 1 prior chemotherapy (excluding prior neo-adjuvant or adjuvant chemotherapy or chemoradiotherapy with curative intent)
* Any toxicity related to prior EGFR inhibitor treatment must have resolved to Grade 1 or less
* Central laboratory confirmation of the presence of the T790M mutation in tumor tissue in Cohort A and the presence or absence of the T790M mutation in tumor tissue in Cohort B. Centrally indeterminate, unknown or invalid specimens are not acceptable. Biopsy material obtained from either primary or metastatic tumor tissue and sent to the central laboratory must be within 60 prior to dosing study drug but following disease progression on the first EGFR TKI
* Measurable disease according to RECIST Version 1.1
* Life expectancy of at least 3 months
* ECOG performance status of 0 to 1
* Minimum Age 18 years (in certain territories, the minimum age requirement may be higher eg age 20 years in Japan and Taiwan)
* Adequate hematological and biological function, confirmed by defined laboratory values
* Written consent on an IRB/IEC-approved Informed Consent Form (ICF) prior to any study specific evaluation

Exclusion Criteria

* Documented evidence of an exon 20 insertion activating mutation in the EGFR gene
* Active second malignancy i.e. patient known to have potentially fatal cancer present for which he/she may be (but not necessarily) currently receiving treatment
* Patients with a history of malignancy that has been completely treated, with no evidence of that cancer currently, are permitted to enrol in the trial provided all chemotherapy was completed greater than 6 months prior and/or bone marrow transplant greater than 2 years prior
* Known pre-existing interstitial lung disease
* Cohort A only: Patients with leptomeningeal carcinomatosis are excluded. Other central nervous system (CNS) metastases are only permitted if treated, asymptomatic, and stable (not requiring steroid for at least 4 weeks prior to the start of study treatment). Cohort B only: Patients with CNS metastases or leptomeningeal carcinomatosis are excluded.
* Treatment with prohibited medications less than or equal to 14 days prior to treatment with rociletinib
* Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication before starting rociletinib
* Prior treatment with rociletinib, or other drugs that target T790M positive mutant EGFR with sparing of wild type EGFR
* Any of the following cardiac abnormalities or history
* Clinically significant abnormal 12-lead ECG, QT interval corrected using Fridericia's method (QTCF) greater than 450 msec
* Inability to measure QT interval on ECG
* Personal or family history of long QT syndrome
* Implantable pacemaker or implantable cardioverter defibrillator
* Resting bradycardia less than 55 beats/min
* Non-study related surgical procedures less than or equal to 7 days prior to administration of rociletinib. In all cases, the patient must be sufficiently recovered and stable before treatment administration
* Females who are pregnant or breastfeeding
* Refusal to use adequate contraception for fertile patients (females and males) while on treatment and for 12 weeks after the last dose of rociletinib
* Presence of any serious or unstable concomitant systemic disorder incompatible with the clinical study
* Any other reason the investigator considers the patient should not participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2014-06-16 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-08-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (91):
- United States (41):
  - UCLA Medical Center, Alhambra, California
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - Saint Jude Heritage Healthcare, Fullerton, California
  - University of California San Diego Moores Cancer Center, La Jolla, California
  - Northridge Hospital Medical Center, Northridge, California
  - Cancer Care Associates, Redondo Beach, California
  - University of California Davis Medical Center, Sacramento, California
  - University of California San Francisco, San Francisco, California
  - Coastal Integrative Cancer Care, San Luis Obispo, California
  - Saint Mary's Regional Cancer Center, Grand Junction, Colorado
  - Rocky Mountain Cancer Centers, LLP, Lone Tree, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Advanced Medical Specialties, Miami, Florida
  - Cleveland Clinic Florida, Weston, Florida
  - Northwestern University Feinberg School of Medicine, Chicago, Illinois
  - University of Illinois Chicago, Chicago, Illinois
  - Illinois Cancer Specialists, Niles, Illinois
  - Beth Israel Comprehensive Cancer Center, Boston, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Minnesota Oncology Hematology, P.A, Minneapolis, Minnesota
  - Mayo Clinic - Rochester, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - New York Oncology Hematology, PC, Latham, New York
  - University of Rochester, Rochester, New York
  - Montefiore Medical Center, The Bronx, New York
  - University Hospitals of Cleveland, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Texas Oncology P.A., Amarillo, Texas
  - USO - Texas Oncology P.A., Arlington, Texas
  - Texas Oncology-Austin Central, Austin, Texas
  - Texas Oncology-Beaumont, Beaumont, Texas
  - Texas Oncology P.A., Bedford, Texas
  - Texas Oncology P.A., Dallas, Texas
  - Texas Oncology P.A., Flower Mound, Texas
  - The Methodist Hospital, Houston, Texas
  - Texas Oncology - Plano East, Plano, Texas
  - Virginia Cancer Specialists, Fairfax, Virginia
  - Northwest Cancer Specialists, P.C., Vancouver, Washington
  - Yakima Valley Memorial Hospital, North Star Lodge, Yakima, Washington
- Australia (4):
  - Icon Cancer Centre, South Brisbane, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Flinders Medical Centre, Bedford Park, South Australia
- Princess Margaret Hospital, Toronto, Ontario, Canada
- France (7):
  - Centre Hospitalier Lyon Sud, Pierre Bénité Cedex, Auvergne-Rhône-Alpes
  - Centre Hospitalier Regional Universitaire (CHRU) de Besancon - L'Hopital Jean Minjoz, Besançon, Franche-comte
  - Institut de Cancérologie de l'Ouest - René Gauducheau, Saint-Herblain, Pays de la Loire Region
  - Centre Hospitalier Universitaire Côte de Nacre, Caen
  - Centre Hospitalier Universitaire Hôpital Nord, Marseille
  - Hôpital Tenon, Paris, Île-de-France Region
  - Institut Gustave Roussy, Villejuif, Île-de-France Region
- Germany (9):
  - Asklepios Fachkliniken München-Gauting, Gauting, Bavaria
  - Klinikum Innenstadt LMU, München, Bavaria
  - Goethe-Universität Frankfurt am Main, Frankfurt am Main, Hesse
  - Pius Hospital Oldenburg, Oldenburg, Lower Saxony
  - Universitaetsklinikum Bonn - Zentrum fuer Innere Medizin - Medizinische Klinik und Poliklink III, Bonn, North Rhine-Westphalia
  - Universitätsklinikum Köln, Cologne, North Rhine-Westphalia
  - Universitätsklinikum Essen, Essen, North Rhine-Westphalia
  - LungenClinic Großhansdorf GmbH, Großhansdorf, Schleswig-Holstein
  - Evangelische Lungenklinik Berlin, Berlin
- Queen Mary Hospital, Hong Kong, Hong Kong
- Netherlands (2):
  - Antoni van Leeuwenhoek Hospital, Amsterdam, North Holland
  - Vrije Universiteit Medisch Centrum, Amsterdam
- South Korea (10):
  - National Cancer Center, Goyang-si, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon, Gyeonggi-do
  - Chungbuk National University Hospital, Chungju, North Chungcheong
  - Dong-A University Hospital, Busan
  - Inha University Hospital, Incheon
  - Samsung Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Hospital, Seoul
  - Seoul Saint Mary's Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (5):
  - Hospital Universitario Virgen del Rocio, Seville, Sevilla
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital Vall d´Hebrón, Barcelona
  - Hospital Universitario Quirón Dexeus, Barcelona
  - Hospital Universitario La Paz, Madrid
- Centre Hospitalier Universitaire Vaudoise, Lausanne, Canton of Vaud, Switzerland
- Taiwan (5):
  - Taipei Veterans General Hospital, Taipei, Taipei CITY
  - Chang Gung Memorial Hospital Linkou, Taoyuan District, Tao-Yuan
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
- United Kingdom (5):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge, England
  - Guy's and Saint Thomas NHS Foundation Trust, London, Greater London
  - Royal Marsden Hospital, London, Greater London
  - Royal Marsden NHS Trust, Sutton, Surrey
  - University College Hospital, London

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 318 patients were enrolled at 67 study sites in North America, Europe, Asia and Australia. One patient was not included in the Safety Population due to failure of the study site to provide any dosing data in electronic data capture (EDC) before the site was closed.
Groups:
- Rociletinib 625 mg BID T790M+: Rociletinib 625 mg BID in patients with T790M-positive tumor status
- Rociletinib 500 mg BID T790M+: Rociletinib 500 mg BID in patients with T790M-positive tumor status
- Rociletinib 500 mg BID T790M-: Rociletinib 500 mg BID in patients with T790M-negative tumor status
Period: Overall Study
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | Rociletinib 500 mg BID T790M-
Started | 154 | 100 | 63
Completed | 154 | 100 | 63
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | Rociletinib 500 mg BID T790M- | Total
Number analyzed (Participants) | 154 | 100 | 63 | 317
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.8 (10.67) | 65.3 (9.93) | 64.1 (10.01) | 63.8 (10.34)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 69 | 41 | 215
  Male | 49 | 31 | 22 | 102
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 3 | 7
  Not Hispanic or Latino | 131 | 93 | 55 | 279
  Unknown or Not Reported | 21 | 5 | 5 | 31
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 59 | 34 | 32 | 125
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 6 | 5 | 2 | 13
  White | 74 | 58 | 23 | 155
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 14 | 3 | 6 | 23
T790M Status [Count of Participants; unit: Participants]
  T790M Negative | 1 | 0 | 62 | 63
  T790M Positive | 153 | 100 | 0 | 253
  Missing | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) According to RECIST Version 1.1 as Determined by Investigator Assessment
Description: ORR is defined as the percentage of patients with a best overall confirmed response of partial response (PR) or complete response (CR) recorded from the start of the treatment until disease progression. For patients who continued treatment post-progression, the first date of progression was used for the analysis. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions, defined by and assessed as: Complete Response (CR), is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial Response (PR), at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter.
Time Frame: Cycle 1 Day 1 to End of Treatment, up to approximately 57 months.
Population: Investigator Tumor Evaluable Population - defined as all patients who received at least 1 dose of rociletinib, have at least 1 measureable tumor lesion at baseline, and have at least 1 post-baseline tumor assessment as determined by the investigator.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | Rociletinib 500 mg BID T790M-
Number analyzed (Participants) | 153 | 97 | 61
percentage of participants | 34.6 [27.1 to 42.7] | 34.0 [24.7 to 44.3] | 18.0 [9.4 to 30.0]

2. Secondary Outcome: Duration of Response (DOR) in T790M Positive Patients According to RECIST Version 1.1 as Determined by Investigator Assessment
Description: DOR in patients with a T790M mutation (determined by central lab) with confirmed response per investigator. The DOR for complete response (CR) and partial response (PR) was measured from the date that any of these best responses is first recorded until the first date that progressive disease (PD) is objectively documented. For patients who continue treatment post-progression, the first date of progression was used for the analysis.
Time Frame: From Cycle 1 Day 1 until disease progression or end of treatment, whichever came first, assessed up to 54 months
Population: Centrally-confirmed T790M-positive subset of the Investigator Tumor Evaluable Population - defined as all patients who received at least 1 dose of rociletinib, have at least 1 measureable tumor lesion at baseline, and have at least 1 post-baseline tumor assessment as determined by the investigator.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- All T790M+: All Rociletinib 500 mg BID and 625 mg BID patients with T790M-positive tumor status
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | All T790M+
Number analyzed (Participants) | 53 | 33 | 86
months | 7.4 [5.5 to 9.4] | 9.1 [5.6 to 13.0] | 7.6 [7.3 to 9.4]

3. Secondary Outcome: Disease Control Rate (DCR) by RECIST v1.1 as Determined by Investigator Assessment
Description: DCR is defined as the percentage of patients who have achieved CR, PR, and SD lasting at least 12 weeks. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions, defined by and assessed as: Complete Response (CR), is disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to < 10 mm. Partial Response (PR), at least a 30% decrease in the sum of the longest diameter of target lesions, taking as reference the baseline sum of longest diameter. Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for progressive disease (PD), taking as reference the smallest sum longest diameter since the treatment started.
Time Frame: From Cycle 1 Day 1 until disease progression or end of treatment, whichever came first, assessed up to 57 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | Rociletinib 500 mg BID T790M-
Number analyzed (Participants) | 153 | 97 | 61
percentage of patients | 67.3 [59.3 to 74.7] | 76.3 [66.6 to 84.3] | 59.0 [45.7 to 71.4]

4. Secondary Outcome: Progression-free Survival (PFS) in T790M Positive Patients by RECIST v1.1 as Determined by Investigator Assessment
Description: PFS was calculated as 1+ the number of days from the first dose of study drug to documented radiographic progression or death due to any cause, whichever occurs first. Patients without a documented event of radiographic progression were censored on the date of their last adequate tumor assessment (i.e., radiologic assessment) or date of first dose of study drug if no tumor assessments were performed. For patients who continued treatment post-progression, the first date of progression was used for the analysis of PFS. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), at least a 20% increase in the sum of the longest diameter of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions is also considered progression.
Time Frame: From Cycle 1 Day 1 until disease progression or end of treatment, whichever came first, assessed up to 57 months
Population: Centrally-confirmed T790M-positive subset of the Intent-to-treat (ITT) population defined as all patients who received at least 1 dose of rociletinib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | All T790M+
Number analyzed (Participants) | 154 | 100 | 254
months | 5.5 [4.0 to 6.7] | 5.9 [5.3 to 8.3] | 5.5 [5.3 to 7.2]

5. Secondary Outcome: Overall Survival (OS) Determined by Investigator Assessment
Description: OS was calculated as 1+ the number of days from the first dose of study drug to death due to any cause. Patients without a documented date of death will be censored on the date the patient was last known to be alive.
Time Frame: Cycle 1 Day 1 to date of death, assessed up to 57 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | All T790M+
Number analyzed (Participants) | 154 | 100 | 254
months | 18.8 [15.2 to NA] — There are an insufficient number of participants with events. | 29.8 [26.2 to NA] — There are an insufficient number of participants with events. | 23.7 [17.7 to 40.6]

6. Secondary Outcome: Change From Baseline to Cycles 5, 10 and End of Treatment (EOT) in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Cancer (EORTC QLQ-C30) Global Health Status Quality of Life Scale
Description: EORTC QLC-C30 is a 30-item questionnaire to assess the quality of life in cancer patients. EORTC QLQ-C30 includes functional scales (physical, role, cognitive, emotional, social), global health status, symptom scales (fatigue, pain, nausea/vomiting), and other (dyspnoea, appetite loss, insomnia, constipation/diarrhea, financial difficulties). Most questions used 4-point scale (1 'Not at All' to 4 'Very Much'); two used 7-point scale (1 'Very Poor' to 7 'Excellent'). Scores are averaged, and transformed to 0-100 scale; higher score = better quality of life.
Time Frame: Baseline (Day 0), Months 5, 10 and EOT
Population: Safety population - defined as all patients who received at least 1 dose of rociletinib.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | Rociletinib 500 mg BID T790M-
Number analyzed (Participants) | 154 | 100 | 63
units on a scale
  Baseline (Day 0): number analyzed (Participants) | 154 | 99 | 63
  Baseline (Day 0) | 62.18 (22.245) | 59.76 (22.495) | 54.63 (24.629)
  Cycle 5 (approximately month 5): number analyzed (Participants) | 101 | 60 | 33
  Cycle 5 (approximately month 5) | -2.48 (22.470) | -0.56 (23.763) | 5.56 (28.842)
  Cycle 10 (approximately month 10): number analyzed (Participants) | 49 | 35 | 14
  Cycle 10 (approximately month 10) | -2.21 (22.294) | -3.81 (21.422) | 3.57 (23.956)
  End of Treatment: number analyzed (Participants) | 38 | 19 | 16
  End of Treatment | -4.82 (23.381) | -9.65 (18.481) | -10.42 (35.158)

7. Secondary Outcome: Change From Baseline to Cycles 5, 10 and End of Treatment (EOT) in Dermatology Life Quality Index (DLQI)
Description: Dermatology Life Quality Index (DLQI) score is a participant-reported outcome consisting of a set of 10 questions regarding the degree to which the participant's skin has affected certain behaviors and quality of life over the last week. Responses to each are: very much (score of 3), a lot, a little, or not at all (score of 0). The DLQI score ranges from 0 (best) to 30 (worst); the higher the score, the more quality of life is impaired.
Time Frame: Baseline (Day 0), Months 5, 10 and EOT
Population: Safety population - defined as all patients who received at least 1 dose of rociletinib.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | Rociletinib 500 mg BID T790M-
Number analyzed (Participants) | 154 | 100 | 63
units on a scale
  Baseline (Day 0): number analyzed (Participants) | 152 | 97 | 62
  Baseline (Day 0) | 2.10 (3.408) | 2.42 (4.706) | 2.74 (4.763)
  Cycle 5 (approximately month 5): number analyzed (Participants) | 97 | 58 | 32
  Cycle 5 (approximately month 5) | -0.82 (3.240) | -1.29 (3.499) | -1.63 (3.731)
  Cycle 10 (approximately month 10): number analyzed (Participants) | 49 | 36 | 14
  Cycle 10 (approximately month 10) | -1.02 (2.810) | -1.64 (3.531) | -0.79 (2.751)
  End of Treatment: number analyzed (Participants) | 35 | 18 | 14
  End of Treatment | -0.77 (3.191) | -0.22 (2.157) | -1.14 (4.204)

8. Secondary Outcome: Change From Baseline to Cycles 5, 10 and End of Treatment (EOT) in EORTC QLQ-LC-13 Alopecia Scale
Description: EORTC QLQ-LC13 is the lung cancer module of EORTC QLQ-C30 and includes questions specific to the disease associated symptoms (dyspnea, cough, hemoptysis, and site specific pain), treatment-related symptoms (sore mouth, dysphagia, neuropathy and alopecia), and analgesic use of lung cancer patients. The scale was transformed to a range of 0 to 100 using standard EORTC algorithm. Higher score indicates worse symptoms.
Time Frame: Baseline (Day 0), Months 5, 10 and EOT
Population: Safety population - defined as all patients who received at least 1 dose of rociletinib.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | Rociletinib 500 mg BID T790M-
Number analyzed (Participants) | 154 | 100 | 63
units on a scale
  Baseline (Day 0): number analyzed (Participants) | 154 | 99 | 63
  Baseline (Day 0) | 9.96 (21.264) | 9.43 (20.779) | 19.05 (29.154)
  Cycle 5 (approximately month 5): number analyzed (Participants) | 101 | 62 | 33
  Cycle 5 (approximately month 5) | -4.62 (27.499) | -2.69 (27.855) | -10.10 (19.516)
  Cycle 10 (approximately month 10): number analyzed (Participants) | 50 | 35 | 13
  Cycle 10 (approximately month 10) | -2.00 (21.728) | -6.67 (25.309) | -2.56 (21.350)
  End of Treatment: number analyzed (Participants) | 37 | 19 | 15
  End of Treatment | 4.50 (33.483) | 3.51 (44.298) | 0.00 (39.841)

9. Secondary Outcome: Change From Baseline to Cycles 5, 10 and End of Treatment (EOT) in EORTC QLQ-LC-13 Coughing Scale
Description: as for outcome 8
Time Frame: Baseline (Day 0), Months 5, 10 and EOT
Population: Safety population - defined as all patients who received at least 1 dose of rociletinib.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | Rociletinib 500 mg BID T790M-
Number analyzed (Participants) | 154 | 100 | 63
units on a scale
  Baseline (Day 0): number analyzed (Participants) | 154 | 99 | 63
  Baseline (Day 0) | 33.12 (26.540) | 29.97 (25.862) | 38.62 (23.346)
  Cycle 5 (approximately month 5): number analyzed (Participants) | 101 | 61 | 33
  Cycle 5 (approximately month 5) | -7.92 (26.728) | -9.29 (26.619) | -12.12 (27.409)
  Cycle 10 (approximately month 10): number analyzed (Participants) | 50 | 35 | 13
  Cycle 10 (approximately month 10) | -6.67 (23.328) | -17.14 (30.648) | 2.56 (21.350)
  End of Treatment: number analyzed (Participants) | 37 | 19 | 15
  End of Treatment | -5.41 (27.793) | 0.00 (36.851) | 6.67 (25.820)

10. Secondary Outcome: Change From Baseline to Cycles 5, 10 and End of Treatment (EOT) in EORTC QLQ-LC-13 Dysphagia Scale
Description: as for outcome 8
Time Frame: Baseline (Day 0), Months 5, 10 and EOT
Population: Safety population - defined as all patients who received at least 1 dose of rociletinib.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | Rociletinib 500 mg BID T790M-
Number analyzed (Participants) | 154 | 100 | 63
units on a scale
  Baseline (Day 0): number analyzed (Participants) | 154 | 99 | 63
  Baseline (Day 0) | 5.19 (15.306) | 7.41 (17.532) | 5.82 (17.495)
  Cycle 5 (approximately month 5): number analyzed (Participants) | 101 | 62 | 33
  Cycle 5 (approximately month 5) | 1.65 (12.803) | -0.54 (17.589) | 7.07 (21.663)
  Cycle 10 (approximately month 10): number analyzed (Participants) | 51 | 35 | 13
  Cycle 10 (approximately month 10) | -3.27 (13.752) | -3.81 (15.700) | 2.56 (9.245)
  End of Treatment: number analyzed (Participants) | 37 | 18 | 15
  End of Treatment | 3.60 (17.184) | 7.41 (31.427) | 6.67 (28.730)

11. Secondary Outcome: Change From Baseline to Cycles 5, 10 and End of Treatment (EOT) in EORTC QLQ-LC-13 Dyspnoea Scale
Description: as for outcome 8
Time Frame: Baseline (Day 0), Months 5, 10 and EOT
Population: Safety population - defined as all patients who received at least 1 dose of rociletinib.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | Rociletinib 500 mg BID T790M-
Number analyzed (Participants) | 154 | 100 | 63
units on a scale
  Baseline (Day 0): number analyzed (Participants) | 154 | 99 | 63
  Baseline (Day 0) | 21.79 (21.554) | 22.56 (21.441) | 30.34 (26.415)
  Cycle 5 (approximately month 5): number analyzed (Participants) | 101 | 62 | 33
  Cycle 5 (approximately month 5) | 6.11 (21.681) | -1.25 (18.777) | -3.70 (23.516)
  Cycle 10 (approximately month 10): number analyzed (Participants) | 51 | 35 | 13
  Cycle 10 (approximately month 10) | 2.83 (19.606) | 1.90 (14.879) | 6.84 (22.923)
  End of Treatment: number analyzed (Participants) | 37 | 19 | 15
  End of Treatment | 8.41 (22.892) | 8.77 (18.362) | 0.00 (28.172)

12. Secondary Outcome: Change From Baseline to Cycles 5, 10 and End of Treatment (EOT) in EORTC QLQ-LC-13 Haemoptysis Scale
Description: as for outcome 8
Time Frame: Baseline (Day 0), Months 5, 10 and EOT
Population: Safety population - defined as all patients who received at least 1 dose of rociletinib.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | Rociletinib 500 mg BID T790M-
Number analyzed (Participants) | 154 | 100 | 63
units on a scale
  Baseline (Day 0): number analyzed (Participants) | 154 | 99 | 63
  Baseline (Day 0) | 2.38 (8.613) | 1.68 (11.039) | 4.76 (13.194)
  Cycle 5 (approximately month 5): number analyzed (Participants) | 101 | 62 | 32
  Cycle 5 (approximately month 5) | -1.98 (7.919) | -1.61 (9.404) | -5.21 (14.930)
  Cycle 10 (approximately month 10): number analyzed (Participants) | 51 | 35 | 13
  Cycle 10 (approximately month 10) | -0.65 (8.138) | -0.95 (5.634) | -5.13 (18.490)
  End of Treatment: number analyzed (Participants) | 37 | 19 | 15
  End of Treatment | -0.90 (12.389) | 0.00 (0.000) | -2.22 (8.607)

13. Secondary Outcome: Change From Baseline to Cycles 5, 10 and End of Treatment (EOT) in EORTC QLQ-LC-13 Pain in Arm or Shoulder Scale
Description: as for outcome 8
Time Frame: Baseline (Day 0), Months 5, 10 and EOT
Population: Safety population - defined as all patients who received at least 1 dose of rociletinib.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | Rociletinib 500 mg BID T790M-
Number analyzed (Participants) | 154 | 100 | 63
units on a scale
  Baseline (Day 0): number analyzed (Participants) | 154 | 98 | 61
  Baseline (Day 0) | 19.91 (26.271) | 16.67 (26.325) | 28.42 (34.338)
  Cycle 5 (approximately month 5): number analyzed (Participants) | 101 | 62 | 32
  Cycle 5 (approximately month 5) | -5.94 (32.110) | -2.69 (25.819) | -7.29 (35.655)
  Cycle 10 (approximately month 10): number analyzed (Participants) | 51 | 35 | 12
  Cycle 10 (approximately month 10) | -1.31 (31.242) | -2.86 (27.262) | 8.33 (28.868)
  End of Treatment: number analyzed (Participants) | 37 | 19 | 15
  End of Treatment | 5.41 (29.932) | 0.00 (35.136) | 4.44 (33.014)

14. Secondary Outcome: Change From Baseline to Cycles 5, 10 and End of Treatment (EOT) in EORTC QLQ-LC-13 Pain in Chest Scale
Description: as for outcome 8
Time Frame: Baseline (Day 0), Months 5, 10 and EOT
Population: Safety population - defined as all patients who received at least 1 dose of rociletinib.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | Rociletinib 500 mg BID T790M-
Number analyzed (Participants) | 154 | 100 | 63
units on a scale
  Baseline (Day 0): number analyzed (Participants) | 154 | 99 | 63
  Baseline (Day 0) | 19.91 (25.429) | 12.79 (22.691) | 25.40 (32.635)
  Cycle 5 (approximately month 5): number analyzed (Participants) | 101 | 62 | 33
  Cycle 5 (approximately month 5) | -4.62 (25.399) | -5.38 (20.194) | -8.08 (28.904)
  Cycle 10 (approximately month 10): number analyzed (Participants) | 51 | 34 | 13
  Cycle 10 (approximately month 10) | -3.27 (24.272) | -6.86 (19.728) | 2.56 (39.585)
  End of Treatment: number analyzed (Participants) | 37 | 19 | 15
  End of Treatment | 1.80 (34.198) | 7.02 (13.962) | -4.44 (30.516)

15. Secondary Outcome: Change From Baseline to Cycles 5, 10 and End of Treatment (EOT) in EORTC QLQ-LC-13 Medicine for Pain Scale
Description: as for outcome 8
Time Frame: Baseline (Day 0), Months 5, 10 and EOT
Population: Safety population - defined as all patients who received at least 1 dose of rociletinib.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | Rociletinib 500 mg BID T790M-
Number analyzed (Participants) | 154 | 100 | 63
units on a scale
  Baseline (Day 0): number analyzed (Participants) | 86 | 50 | 42
  Baseline (Day 0) | 60.47 (27.302) | 66.67 (27.766) | 53.17 (23.350)
  Cycle 5 (approximately month 5): number analyzed (Participants) | 30 | 15 | 14
  Cycle 5 (approximately month 5) | 6.67 (35.450) | 8.89 (23.458) | -4.76 (36.648)
  Cycle 10 (approximately month 10): number analyzed (Participants) | 14 | 8 | 3
  Cycle 10 (approximately month 10) | 4.76 (12.105) | -4.17 (27.817) | 22.22 (19.245)
  End of Treatment: number analyzed (Participants) | 17 | 8 | 6
  End of Treatment | 3.92 (20.008) | 0.00 (30.861) | -5.56 (38.968)

16. Secondary Outcome: Change From Baseline to Cycles 5, 10 and End of Treatment (EOT) in EORTC QLQ-LC-13 Pain in Other Parts Scale
Description: as for outcome 8
Time Frame: Baseline (Day 0), Months 5, 10 and EOT
Population: Safety population - defined as all patients who received at least 1 dose of rociletinib.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | Rociletinib 500 mg BID T790M-
Number analyzed (Participants) | 154 | 100 | 63
units on a scale
  Baseline (Day 0): number analyzed (Participants) | 149 | 97 | 61
  Baseline (Day 0) | 28.41 (30.848) | 30.58 (33.219) | 31.69 (29.456)
  Cycle 5 (approximately month 5): number analyzed (Participants) | 95 | 59 | 30
  Cycle 5 (approximately month 5) | 2.46 (34.464) | -1.13 (29.664) | -7.78 (33.543)
  Cycle 10 (approximately month 10): number analyzed (Participants) | 48 | 35 | 12
  Cycle 10 (approximately month 10) | -3.47 (28.550) | -6.67 (31.102) | -2.78 (22.285)
  End of Treatment: number analyzed (Participants) | 34 | 17 | 15
  End of Treatment | 20.59 (31.798) | 0.00 (26.352) | 6.67 (44.006)

17. Secondary Outcome: Change From Baseline to Cycles 5, 10 and End of Treatment (EOT) in EORTC QLQ-LC-13 Peripheral Neuropathy Scale
Description: as for outcome 8
Time Frame: Baseline (Day 0), Months 5, 10 and EOT
Population: Safety population - defined as all patients who received at least 1 dose of rociletinib.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | Rociletinib 500 mg BID T790M-
Number analyzed (Participants) | 154 | 100 | 63
units on a scale
  Baseline (Day 0): number analyzed (Participants) | 154 | 99 | 62
  Baseline (Day 0) | 11.90 (22.117) | 6.40 (17.611) | 17.20 (29.409)
  Cycle 5 (approximately month 5): number analyzed (Participants) | 101 | 62 | 32
  Cycle 5 (approximately month 5) | 0.00 (25.386) | 3.76 (23.458) | 4.17 (31.395)
  Cycle 10 (approximately month 10): number analyzed (Participants) | 51 | 35 | 12
  Cycle 10 (approximately month 10) | 4.58 (25.837) | 2.86 (18.737) | 0.00 (20.101)
  End of Treatment: number analyzed (Participants) | 37 | 19 | 15
  End of Treatment | 2.70 (21.341) | 7.02 (26.244) | 2.22 (15.258)

18. Secondary Outcome: Change From Baseline to Cycles 5, 10 and End of Treatment (EOT) in EORTC QLQ-LC-13 Sore Mouth Scale
Description: as for outcome 8
Time Frame: Baseline (Day 0), Months 5, 10 and EOT
Population: Safety population - defined as all patients who received at least 1 dose of rociletinib.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | Rociletinib 500 mg BID T790M-
Number analyzed (Participants) | 154 | 100 | 63
units on a scale
  Baseline (Day 0): number analyzed (Participants) | 154 | 99 | 63
  Baseline (Day 0) | 5.19 (13.273) | 7.41 (17.532) | 10.58 (21.440)
  Cycle 5 (approximately month 5): number analyzed (Participants) | 101 | 61 | 33
  Cycle 5 (approximately month 5) | 1.98 (18.149) | -2.19 (21.832) | -2.02 (27.562)
  Cycle 10 (approximately month 10): number analyzed (Participants) | 51 | 35 | 13
  Cycle 10 (approximately month 10) | 0.65 (19.425) | -1.90 (24.176) | 2.56 (21.350)
  End of Treatment: number analyzed (Participants) | 37 | 19 | 15
  End of Treatment | 4.50 (21.026) | 12.28 (29.836) | 2.22 (36.659)

19. Secondary Outcome: Population PK (POPPK) and Exposure-Response (ER) Analysis of Rociletinib
Description: Sparse blood sampling for POPPK and ER analyses in all patients treated with rociletinib.
Time Frame: Every 4 weeks for approximately 6 months (Day 1 of Cycles 2 to 7 inclusive)
Population: Population PK (PPK) and exposure-response (ER) analysis were listed as a secondary objective. These analyses were conducted based on pooled data from multiple rociletinib trials (including TIGER2), thus no PPK or ER report was generated specifically for this study.
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | Rociletinib 500 mg BID T790M-
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the date of first dose of study drug and within 28 days after last dose of study drug, or up to approximately 62 months. In addition, study procedure-related AEs that occurred after signing of the informed consent form and before first dose of study drug were expected to be reported.
Arm/Group | Rociletinib 625 mg BID T790M+ | Rociletinib 500 mg BID T790M+ | Rociletinib 500 mg BID T790M-
All-Cause Mortality (participants affected / at risk) | 27/154 | 7/100 | 9/63
Serious Adverse Events (participants affected / at risk) | 77/154 | 48/100 | 34/63
Other Adverse Events (participants affected / at risk) | 153/154 | 100/100 | 63/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rociletinib 625 mg BID T790M+ (N=154) | Rociletinib 500 mg BID T790M+ (N=100) | Rociletinib 500 mg BID T790M- (N=63)
Anemia (Blood and lymphatic system disorders) | 3 | 0 | 1
Lymphadenitis (Blood and lymphatic system disorders) | 1 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 0 | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 2
Bradycardia (Cardiac disorders) | 2 | 0 | 0
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 2 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 1 | 0 | 0
Angle closure glaucoma (Eye disorders) | 0 | 2 | 0
Cataract (Eye disorders) | 2 | 2 | 4
Diplopia (Eye disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 0
Duodenal ulcer (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 0 | 1 | 0
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 6 | 2 | 2
Pancreatitis (Gastrointestinal disorders) | 5 | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 4 | 3 | 3
Chest pain (General disorders) | 2 | 2 | 0
Death (General disorders) | 1 | 0 | 0
Euthanasia (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 0 | 2 | 0
Malaise (General disorders) | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Oedema (General disorders) | 0 | 0 | 1
Oedema peripheral (General disorders) | 0 | 0 | 1
Peripheral swelling (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 1 | 3 | 1
Sudden death (General disorders) | 0 | 0 | 1
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 2
Cholecystitis acute (Hepatobiliary disorders) | 1 | 2 | 0
Gallbladder obstruction (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 1 | 0
Hepatitis (Hepatobiliary disorders) | 1 | 0 | 0
Biliary tract infection (Infections and infestations) | 1 | 0 | 0
Cellulitis (Infections and infestations) | 1 | 0 | 0
Clostridium difficile infection (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Listeria sepsis (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 2
Pneumonia (Infections and infestations) | 3 | 5 | 2
Pneumonia bacterial (Infections and infestations) | 0 | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 2 | 0
Sepsis (Infections and infestations) | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 3 | 0
Postoperative ileus (Injury, poisoning and procedural complications) | 0 | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0 | 2
Electrocardiogram QT prolonged (Investigations) | 2 | 0 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0
Transaminases increased (Investigations) | 1 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 2 | 0
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 10 | 6 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 0
Bursitis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 2 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pathological fracture (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 23 | 4 | 7
Malignant pleural effusion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Myelodysplastic syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 1
Leukoencephalopathy (Nervous system disorders) | 1 | 0 | 0
Partial seizures (Nervous system disorders) | 1 | 0 | 0
Seizure (Nervous system disorders) | 2 | 1 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 2 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Bladder perforation (Renal and urinary disorders) | 1 | 0 | 0
Cystitis interstitial (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 1
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 4 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 0
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 0 | 0
Embolism (Vascular disorders) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Shock haemorrhagic (Vascular disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rociletinib 625 mg BID T790M+ (N=154) | Rociletinib 500 mg BID T790M+ (N=100) | Rociletinib 500 mg BID T790M- (N=63)
Anaemia (Blood and lymphatic system disorders) | 32 | 13 | 10
Neutropenia (Blood and lymphatic system disorders) | 3 | 5 | 2
Thromobcytopenia (Blood and lymphatic system disorders) | 11 | 1 | 1
Cataract (Eye disorders) | 28 | 18 | 7
Vision blurred (Eye disorders) | 7 | 8 | 2
Abdominal pain (Gastrointestinal disorders) | 24 | 15 | 6
Abdominal pain upper (Gastrointestinal disorders) | 18 | 9 | 1
Constipation (Gastrointestinal disorders) | 38 | 35 | 21
Diarrhoea (Gastrointestinal disorders) | 91 | 59 | 30
Dry mouth (Gastrointestinal disorders) | 18 | 13 | 2
Dyspepsia (Gastrointestinal disorders) | 13 | 4 | 7
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 16 | 8 | 5
Mouth ulceration (Gastrointestinal disorders) | 2 | 2 | 5
Nausea (Gastrointestinal disorders) | 86 | 58 | 31
Stomatitis (Gastrointestinal disorders) | 9 | 5 | 1
Vomiting (Gastrointestinal disorders) | 62 | 35 | 21
Asthenia (General disorders) | 19 | 6 | 6
Chest pain (General disorders) | 11 | 13 | 3
Fatigue (General disorders) | 57 | 48 | 29
Influenza like illness (General disorders) | 8 | 5 | 2
Malaise (General disorders) | 4 | 2 | 4
Mucosal inflammation (General disorders) | 6 | 7 | 3
Non-cardiac chest pain (General disorders) | 8 | 1 | 2
Oedema peripheral (General disorders) | 16 | 6 | 8
Pyrexia (General disorders) | 21 | 11 | 5
Paronychia (Infections and infestations) | 2 | 5 | 0
Pneumonia (Infections and infestations) | 7 | 5 | 5
Upper respiratory tract infection (Infections and infestations) | 13 | 8 | 4
Urinary tract infection (Infections and infestations) | 22 | 15 | 6
Alanine aminotransferase increased (Investigations) | 21 | 9 | 6
Aspartate aminotransferase increased (Investigations) | 18 | 5 | 5
Blood alkaline phosphatase increased (Investigations) | 10 | 6 | 4
Blood bilirubin increased (Investigations) | 15 | 3 | 2
Blood creatinine increased (Investigations) | 12 | 7 | 5
Electrocardiogram QT prolonged (Investigations) | 62 | 29 | 19
Platelet count decreased (Investigations) | 6 | 2 | 4
Weight decreased (Investigations) | 43 | 28 | 15
Decreased appetite (Metabolism and nutrition disorders) | 62 | 42 | 25
Dehydration (Metabolism and nutrition disorders) | 16 | 5 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 97 | 64 | 33
Hypoalbuminaemia (Metabolism and nutrition disorders) | 8 | 3 | 3
Hypokalaemia (Metabolism and nutrition disorders) | 18 | 9 | 8
Hypomagnesaemia (Metabolism and nutrition disorders) | 12 | 7 | 3
Hyponatraemia (Metabolism and nutrition disorders) | 8 | 8 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 22 | 18 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 19 | 9
Muscle spasms (Musculoskeletal and connective tissue disorders) | 35 | 23 | 10
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 11 | 7 | 4
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 13 | 7 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 15 | 4 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 5 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8 | 7 | 3
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 27 | 7 | 9
Dizziness (Nervous system disorders) | 21 | 18 | 7
Dysgeusia (Nervous system disorders) | 10 | 9 | 5
Headache (Nervous system disorders) | 45 | 19 | 14
Lethargy (Nervous system disorders) | 3 | 2 | 4
Anxiety (Psychiatric disorders) | 7 | 4 | 4
Confusional state (Psychiatric disorders) | 8 | 3 | 2
Depression (Psychiatric disorders) | 5 | 6 | 3
Insomnia (Psychiatric disorders) | 13 | 10 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 35 | 25 | 18
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 2 | 6 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 28 | 24 | 15
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 5 | 6 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 4 | 0 | 4
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 7 | 6 | 6
Productive cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 4
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 11 | 8 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 8 | 5 | 7
Rash (Skin and subcutaneous tissue disorders) | 9 | 9 | 2
Hypertension (Vascular disorders) | 9 | 4 | 3
Hypotension (Vascular disorders) | 5 | 5 | 0
Abdominal distension (Gastrointestinal disorders) | 6 | 6 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
All parties agree to submit all manuscripts or abstracts to all other parties 30 days prior to submission. This will enable all parties to protect proprietary information and to provide comments based on information that may not yet be available to other parties. The sponsor may request a delay in publication if there are important intellectual property concerns relating to publication, but does not have the right to suppress publication of the study results indefinitely.

DOCUMENTS (2):
  • Study Protocol (2016-08-16): https://cdn.clinicaltrials.gov/large-docs/90/NCT02147990/Prot_000.pdf
  • Statistical Analysis Plan (2015-06-12): https://cdn.clinicaltrials.gov/large-docs/90/NCT02147990/SAP_001.pdf